CLINICAL TRIAL: NCT04513873
Title: The Effect Of Diverting The Children's Attention To A Different Point During Phlebotomy On Pain And Anxiety
Brief Title: The Effect Of Diverting The Children's Attention To A Different Point During Phlebotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeliz Ciğerci, Assistant Professor PhD, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/37
Record Dates: First submitted 2020-08-08; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Pain and Anxiety of Children During Phlebotomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equipment Intervention Group (Experimental): The intervention group had equipment that looks like a blood tube in front of them during the blood collection process to divert their attention from the blood collection process to the equipment. This equipment was with a fixed arm on the right and a moving arm on the left with a total height of 80 cm as well as a red light-emitting diode(LED) to stimulate the blood collection. It had some answers to common questions of parents as well as the key concerns of the children like " Will it hurt me?". The equipment was made a musical device by loading the most popular children's songs into its database.
  Interventions: Device: Equipment to divert the focus of children
- No Intervention Group (No Intervention): Standard blood collection procedures were applied to the control group.

INTERVENTIONS:
Device: Equipment to divert the focus of children — The equipment was placed in an area where the children would be able to see easily during the blood collection process. It was turned on as soon as the children sat on to the chair where the process would take place to divert the focus of the children at the equipment.
  Arms: Equipment Intervention Group

SUMMARY:
This study aimed to investigate the effect of diverting the children's attention to a different point during phlebotomy which is an invasive procedure with acute pain. This is a randomized controlled experimental study. The study was conducted with two groups: the intervention group (n=127) and the control group (n=129). The control group was applied to standard phlebotomy procedures. In contrast, the intervention group had a piece of equipment that looks like a blood tube in front of them during the phlebotomy process to divert their attention from the phlebotomy process to the equipment.

DETAILED DESCRIPTION:
The equipment used for the intervention group was designed and developed by the researchers with the project support of TÜBİTAK BİDEB 2209A in 2016. It is an equipment that looks like a blood tube with a fixed arm on the right and a moving arm on the left with a total height of 80 cm. It has some answers to common questions of parents as well as the key concerns of the children " Will it hurt me?"

ELIGIBILITY:
Inclusion Criteria:

* making a request for the phlebotomy
* being in the 7-12 age group
* having the consent of the parent
* willing to participate in the research
* with the history of invasive procedure
* not using any medication with analgesic effect in the last 12 hours
* without any communication barriers of either child or the parent
* with a normal level of consciousness during the process
* without the history of passing out during the phlebotomy

Exclusion Criteria:

* not being in the 7-12 age group
* not having the consent of the parent
* not willing to participate in the research
* without the history of invasive procedure
* had medication with analgesic effect in the last 12 hours
* with communication barriers of either child or the parent
* with an abnormal level of consciousness during the process
* with the history of passing out during the phlebotomy

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Assessment of Children's Anxiety Level Change | Twice ( Immediately after the procedure and 14 days after the procedure)
  Children's Fear Scale is an instrument with five different face images changing from neutral (0= no fear) to most scared (4= with the most fear) to evaluate the scare level of the children during the procedure.

SECONDARY OUTCOMES:
Revised Face Pain Scale (FPS-R) | Twice ( During the procedure and 5-10 minutes after the procedure)
  The FPS-R is a scale to measure how children feel in their inner world than how their faces look. It is designed on the widely accepted 0-to-10 metric according to the chosen face. "0" equals "No pain" and "10" equals "Very much pain."

CONTACTS AND LOCATIONS:
Locations (1):
- Manavgat State Hospital, Antalya, Manavgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No